CLINICAL TRIAL: NCT02059460
Title: Perioperative Evaluation of Terlipressin Infusion During Living Donor Liver Transplantation on Incidence of Acute Kidney
Acronym: Terli-NGAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Liver Institute, Egypt (Other)
Collaborators: Dr. Mohamed Helmi Ibrahim Afifi (Unknown); Dr. Khaled Ahmed Yassen (Unknown); Dr. Khalid Mousa Abouelenain (Unknown); Dr. Mohamed Abdelrauf kandil (Unknown); Dr. Ayman Alsebaey Qotb Alghoraieb. (Unknown)
Responsible Party: Principal Investigator, Hanaa Rashed, Assistant lecturer of Anesthesia and Intensive Care, National Liver Institute, Egypt
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Terli-NGAL-111
Record Dates: First submitted 2013-11-10; First posted 2014-02-11 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Acute Kidney Injury; Liver Transplantation; Terlipressin; NGAL
Keywords: Terlipressin; Acute kidney injury; Liver transplantation; NGAL
MeSH Terms: conditions — Acute Kidney Injury | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Terlipressin group (Experimental): Terlipressin group, Terlipressin (Glypressin®, Rentschler biotechnology Gmbh, Erwin, Germany) will be started by continuous infusion at a dose of 1-4 µg/kg/h till day 4 postoperatively
  Interventions: Drug: Terlipressin
- Control group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Terlipressin — Terlipressin (Glypressin®) will be started by continuous infusion at a dose of 1-4 µg/kg/h till day 4 postoperatively
  Other Names: Glypressin
  Arms: Terlipressin group
Drug: placebo
  Arms: Control group

SUMMARY:
To study the impact of intra and post-operative Terlipressin infusion on the occurrence of acute kidney injury after LDLT To investigate perioperative Neutrophil Gelatinase Associated Lipocalin (NGAL) changes and study the effect of Terlipressin on NGAL blood levels

DETAILED DESCRIPTION:
The study will be conducted after approval of the local ethics and research committee of anesthesia, ICU and pain management of both Faculty of Medicine and Liver Institute, Menoufia University, Egypt. This study will be conducted in Anesthesia Department, National Liver Institute hospital on patients undergoing liver transplantation. They will be simply randomized with closed envelopes into two groups. Terlipressin group and Control group. A written informed consent will be taken from every patient.

Inclusion criteria: Adult living donor liver transplant recipients with no preoperative renal dysfunction Exclusion criteria: patients with renal insufficiency defined as serum creatinine > 2 mg/dl and GFR <60 ml/min by isotope scanning of the kidney.

Anesthetic Technique:

All patients will be monitored by electrocardiography, noninvasive and invasive arterial blood pressure, pulse oximetry, capnography, fraction inspired oxygen concentration (FiO2). After preoxygenation, general anesthesia will be induced with Propofol 2 mg/kg IV, Fentanyl 2 µg/kg IV and Rocronium 0.9 mg/kg IV followed by endotracheal intubation and maintenance with a mixture of air, oxygen 50% with Desﬂurane. Mechanical ventilation will be adjusted to maintain end-tidal CO2 between 35-40 mmHg. Central venous line will be inserted for monitoring of central venous pressure (CVP) with ultrasonography guidance.

The esophageal Doppler probe will then be inserted orally and positioned approximately 35-40 cm from the teeth (CardioQTM®, Deltex Medical, Chichester, UK). Normothermia (core temperature > 36°C) will be maintained intraoperatively using forced warming air blanket (Bair Hugger®; Arizant, UK).

After induction of anesthesia patients will be randomly divided into two groups Terlipressin group, Terlipressin (Glypressin®, Rentschler biotechnology Gmbh, Erwin, Germany) will be started by continuous infusion at a dose of 1-4 µg/kg/h till day 4 postoperatively. In the control group, continuous placebo infusion will be started. The Anesthesia team will be kept blind to the contents of the infusion.

Rotetional thromboelastometry [ROTEM] will guide intraoperative blood transfusion protocol as prescribed by the study of Gorlinger K will be followed in both groups. (13) Platelets will be substituted when maximum clot firmness of (MCF EXTEM) <45mm and maximum clot firmness of FIBTEM (MCF FIBTEM) >8mm.

Fresh frozen plasma will be administerd when clot formation time representing extrinsic coagulation pathway (CFT EXTEM) was >240sec. Hematocrite will be kept more than or equal to 25 with packed red blood cells units.

All patients will receive intraoperative methylprednisolone (10 mg/kg). Hemodynamics will be maintained, keeping mean blood pressure above 60 mmHg by fluids and vasoactive drugs.

After surgery, all patients will be transferred to the intensive care unit for controlled mechanical ventilation. The patients will be extubated when hemodynamics are stable, liver graft functions satisfactory, sufficient spontaneous breathing, and core temperature >36°C.

Measured Parameters:

-Evaluation of renal function and injury:

* Serum Cr levels and BUN will be determined preoperatively and then daily up to 5 days after surgery.
* The glomerular ﬁltration rate (GFR) or the nearest approximation of GFR will be calculated from the equation of modiﬁcation of Diet in Renal Disease Study on the basis of obtained serum Cr levels and patient demographics.
* Urine output
* Determination of NGAL Blood samples for the determination of NGAL will be drawn at 3 different time points: immediately after the induction of anesthesia, 2 hours after reperfusion, and 24 hours after reperfusion.

Blood samples will be drawn at the predetermined time points and processed within 2 hours after collection. Serum will be collected and subsequently frozen at -80°Celsius until further analysis -Hemodynamic parameters:

• Heart rate, mean arterial blood pressure [MABP], and CVP, cardiac output (COP), stroke volume (SV), corrected flow time (FTc), systemic vascular resistance (SVR) will be recorded after induction of anesthesia, then every hour during the operation.

Other parameters:

* Anhepatic phase time, warm and cold ischemia time.
* Graft weight , recipient graft body weight ratio.
* Fluid, blood product transfusion.
* Blood glucose level, postoperative complication.
* ICU stay, length of hospital stay.
* 30 days mortality The need for postoperative renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult living donor liver transplant recipients with no preoperative renal dysfunction

Exclusion Criteria:

* patients with renal insufficiency defined as serum creatinine > 2 mg/dl and GFR <60 ml/min by isotope scanning of the kidney.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Development of acute kidney injury | 5 days postoperatuvely
  it is elevation of serum creatinine >1.5 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa S Rashed, MSc, Principal Investigator — National Liver Institute, Egypt
Locations (1):
- National Liver Institute, Shebeen Alkom, Monufia Governorate, Egypt

REFERENCES:
- [Background] Wong F, Nadim MK, Kellum JA, Salerno F, Bellomo R, Gerbes A, Angeli P, Moreau R, Davenport A, Jalan R, Ronco C, Genyk Y, Arroyo V. Working Party proposal for a revised classification system of renal dysfunction in patients with cirrhosis. Gut. 2011 May;60(5):702-9. doi: 10.1136/gut.2010.236133. Epub 2011 Feb 15. PMID 21325171
- [Background] Hong SH, Lee JM, Choi JH, Chung HS, Park JH, Park CS. Perioperative assessment of terlipressin infusion during living donor liver transplantation. J Int Med Res. 2012;40(1):225-36. doi: 10.1177/147323001204000123. PMID 22429362
- [Background] Saner FH, Canbay A, Gerken G, Broelsch CE. Pharmacology, clinical efficacy and safety of terlipressin in esophageal varices bleeding, septic shock and hepatorenal syndrome. Expert Rev Gastroenterol Hepatol. 2007 Dec;1(2):207-17. doi: 10.1586/17474124.1.2.207. PMID 19072411
- [Background] Mishra J, Ma Q, Prada A, Mitsnefes M, Zahedi K, Yang J, Barasch J, Devarajan P. Identification of neutrophil gelatinase-associated lipocalin as a novel early urinary biomarker for ischemic renal injury. J Am Soc Nephrol. 2003 Oct;14(10):2534-43. doi: 10.1097/01.asn.0000088027.54400.c6. PMID 14514731
- [Background] Rostami Z, Nikpoor M, Einollahi B. Urinary Neutrophil Gelatinase Associated Lipocalin (NGAL) for Early Diagnosis of Acute Kidney Injury in Renal Transplant Recipients. Nephrourol Mon. 2013 Spring;5(2):745-52. doi: 10.5812/numonthly.9385. Epub 2013 Mar 30. PMID 23841038
- [Background] Afonso RC, Hidalgo R, Zurstrassen MP, Fonseca LE, Pandullo FL, Rezende MB, Meira-Filho SP, Ferraz-Neto BH. Impact of renal failure on liver transplantation survival. Transplant Proc. 2008 Apr;40(3):808-10. doi: 10.1016/j.transproceed.2008.02.062. PMID 18455024
- [Derived] Kandil MA, Abouelenain KM, Alsebaey A, Rashed HS, Afifi MH, Mahmoud MA, Yassen KA. Impact of terlipressin infusion during and after live donor liver transplantation on incidence of acute kidney injury and neutrophil gelatinase-associated lipocalin serum levels: A randomized controlled trial. Clin Transplant. 2017 Aug;31(8). doi: 10.1111/ctr.13019. Epub 2017 Jun 25. PMID 28564127